CLINICAL TRIAL: NCT06792201
Title: Evaluation of Sarcopenia in Women in Different Stages of Life and in Hormonal Therapy or Not
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SARCWOMEN-20
Record Dates: First submitted 2024-12-30; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Menopause; Hormonal therapy
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intake or not of hormonal therapy of menopause (Other): The study population will be divided into groups according to the intake or not of hormonal therapy of menopause as per normal clinical practice and the menopausal state:
  GROUP A - menopausal patient taking hormone therapy GROUP B - menopausal patient not taking hormone therapy GROUP C - pre-menopausal patients who do not take hormonal products
  Interventions: Diagnostic Test: SARC-F, Handgrip test, Chair stand test

INTERVENTIONS:
Diagnostic Test: SARC-F, Handgrip test, Chair stand test — The SARC-F questionnaire is a simple to use questionnaire consisting of five questions about daily actions.To test the force will be used: Hand-grip test and Chair stand test. The tool used for the hand-grip test is the GRIP-A (Takei). The test is performed on the dominant limb and repeated three times. The position taken by the patient will be: sitting with shoulders and elbows flexed, forearms in neutral position. The Chair stand test measures the time it takes for a patient to get up five times from a sitting position without the help of her upper limbs. The test will be timed.The measurement of lean mass will be carried out by means of a bio impedance meter. This instrument does not measure muscle mass directly but estimates it based on the electrical conductivity of the whole body. Bioimpedance is a method that is easy and safe for the patient to use.
  Other Names: Bioimpedance

SUMMARY:
The three-year interventional study has the following objectives:

The study aims to assess the prevalence of sarcopenia in menopausal women receiving hormone replacement therapy or not compared with pre-menopausal women. The study population will be divided into groups according to the intake or not of hormonal therapy of menopause as per normal clinical practice and the menopausal state:

GROUP A - menopausal patient taking hormone therapy GROUP B - menopausal patient not taking hormone therapy GROUP C - pre-menopausal patients who do not take hormonal products The primary objective is to compare the strength and muscle mass outcomes of HRT in menopausal women compared with those who do not use it and women in pre-menopausal age. Survey methods such as SARC-F, Handgrip test, Chair stand test and bio impedance

DETAILED DESCRIPTION:
The present one-center cross-sectional observational study involves the recruitment of patients attending the O.U. of Gynecology and Pathophysiology of Human Reproduction in menopause who take or do not take hormone replacement therapy at the time of the first visit and women in pre-menopause but similar age group compared to the first group.

Patients will be asked to participate in this study during the outpatient follow-up visit.

The study will involve data collection through consultation of health records.

The objectives of the study will therefore be achieved by analysing certain parameters that can be deduced from the medical records of the subjects in the study:

* Collection of anamnestic (eating habits and sports, pathologies of importance, medication intake, previous surgical interventions, smoking habit, gynecological history).
* Physical examination: calculation of BMI, blood pressure measurement, gynecological examination
* Blood tests (blood count, lipid profile, glycemic, liver, kidney, hormonal status) and urine
* Reports of other visits and specialist examinations performed by the patients brought to view during the visit
* During the visit, the following tests will be proposed:

Questionnaire SARC-F Handgrip test Chair stand test bioimpedance Study population

Inclusion criteria:

* Patients attending the O.U. of Gynecology and Human Reproduction Pathophysiology in menopause who take or do not take hormone replacement therapy at the time of the first visit and women in pre-menopause.
* Patients for whom informed consent has been obtained. Exclusion criteria: no exclusion criteria are provided

Visits and evaluations Visits and assessment scheme Each patient will be invited to participate in this study at the usual outpatient checkup according to current clinical practice. Patients will be free to decide whether or not to participate in the study

Information will be collected from the patients attending the U.O. of Gynecology and Pathophysiology of Human Reproduction in menopause who take or do not take hormone replacement therapy at the time of the first visit and women in pre-menopausemenopause but similar age group compared to the first group.

An estimated sample of 180 subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the O.U. of Gynecology and Pathophysiology of Human Reproduction in menopause who take or do not take hormone replacement therapy at the time of visit as normal clinical practice and women in pre-menopause.

Patients for whom informed consent has been obtained.

Exclusion Criteria:

* no exclusion criteria are provided

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-06-14 (Actual); Primary Completion 2025-06-14 (Estimated); Study Completion 2026-06-14 (Estimated)

PRIMARY OUTCOMES:
Strength and muscle mass outcomes | From enrollment to the end of treatment (1 year)
  The primary objective is to compare the strength and muscle mass outcomes of HRT in menopausal women compared with those who do not use it and women in pre-menopausal age. Survey methods such as SARC-F, Handgrip test, Chair stand test and bio impedance will be used for this purpose.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Meriggiola, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No